CLINICAL TRIAL: NCT02596646
Title: Early Precut Sphincterotomy During ERCP With Difficult Biliary Access (Italian: Esecuzione Del Pre-cut Precoce in Corso di ERCP Con Difficoltosa Incannulazione Della Via Biliare)
Brief Title: Early Precut in Difficult Biliary Cannulation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis recommended terminating the study
Sponsor: Università Vita-Salute San Raffaele (Other)
Collaborators: San Giuseppe Moscati Hospital (Other); Istituti Ospitalieri di Cremona (Other); Valduce Hospital (Other); Papa Giovanni XXIII Hospital (Other); Cardarelli Hospital (Other); Azienda Ospedaliera Universitaria Senese (Other); Maresca Hospital (Other)
Responsible Party: Principal Investigator, Testoni Pier Alberto, Professor, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRECUT PRECOCE/01
Record Dates: First submitted 2015-09-07; First posted 2015-11-04 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Common Bile Duct Diseases
MeSH Terms: conditions — Common Bile Duct Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): Early Precut
  Interventions: Procedure: Early Precut
- Group B (Active Comparator): Prolonged cannulation attempts
  Interventions: Procedure: Prolonged cannulation attempts

INTERVENTIONS:
Procedure: Early Precut — Early precut was performed during ERCP with difficult biliary cannulation
  Arms: Group A
Procedure: Prolonged cannulation attempts — Prolonged cannulation attempts was performed during ERCP with difficult biliary cannulation
  Arms: Group B

SUMMARY:
This study evaluates whether an early precut strategy in cases of difficult biliary cannulation could reduce the incidence of PEP compared with that after prolonged cannulation attempts. Secondary aims are to compare the success of biliary cannulation and complications rates of the two techniques.

DETAILED DESCRIPTION:
In this prospective multicenter randomized clinical trial the investigators assign patients referred for therapeutic biliary ERCP and difficult biliary cannulation (unsuccessful cannulation after 5 minutes) to early precut (group A) or repeated papillary cannulation attempts followed, in case of failure, by late precut (group B). Group A patients undergo precut immediately after randomization ("early precut"), while for group B cannulation attempts are continued for another 10 minutes, after which a precut is done if these fail or there are three unintended additional passages of the guide-wire into the MPD ("delayed precut").

ELIGIBILITY:
Inclusion Criteria:

* 18 to 85 years of age who were scheduled to undergo therapeutic biliary ERCP.

Exclusion Criteria:

* active cholangitis or pancreatitis
* chronic pancreatitis,
* previous sphincterotomy,
* prior gastric surgery,
* coagulopathy,
* severe comorbidity (need for tracheal intubation)
* patients who refused or were unable to give informed consent.
* patients with successful CBD cannulation within 5 minutes of standard attempts and fewer than three passages of the guidewire into the main pancreatic duct (MPD) (arbitrarily defined as "easy CBD cannulation"),
* detection of ampulloma or peri-papillary diverticula during ERCP.

Ages: 18 Years to 85 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Incidence of PEP | 24 hours

SECONDARY OUTCOMES:
Incidence of overall complications | 24 hours
  The incidence of pancreatitis, cholangitis, perforation, bleeding after ERCP was recored. These complications were defined according to the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Pier Alberto Testoni, Professor, Principal Investigator — San Raffaele Hospital
Locations (1):
- San Raffaele Hospital, Milan, Italy